CLINICAL TRIAL: NCT05574660
Title: Influence of High Fat Feeding on Brain and Behaviour in Individuals at Genetic Risk of Obesity
Brief Title: Effect of High-fat/High-sugar Diet on Food Reward Signaling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Max Planck Institute for Metabolism Research (Other)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Marc Tittgemeyer, Prof. Dr., Max Planck Institute for Metabolism Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HF-01
Record Dates: First submitted 2022-10-05; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Behavior, Eating
MeSH Terms: conditions — Feeding Behavior | interventions — Diet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Fat/High-Sugar (HF/HS) Diet (Experimental): Participants randomized to consume an HF/HS yoghurt (40.8 % kcal from fat, 45.6 % kcal from carbohydrates, 13 % kcal from protein of 79.5 total kcal) two times a day for eight weeks in addition to their normal diet.
  Interventions: Dietary Supplement: High-Fat/High-Sugar (HF/HS) Diet
- Low-Fat/Low-Sugar (LF/LS) Diet (Experimental): Participants randomized to consume an LF/LS yoghurt (17.1 % kcal from fat, 29.1 % kcal from carbohydrates, 51.9 % kcal from protein of 78 total kcal) two times a day for eight weeks in addition to their normal diet.
  Interventions: Dietary Supplement: Low-Fat/Low-Sugar (LF/LS) Diet

INTERVENTIONS:
Dietary Supplement: High-Fat/High-Sugar (HF/HS) Diet
  Arms: High-Fat/High-Sugar (HF/HS) Diet
Dietary Supplement: Low-Fat/Low-Sugar (LF/LS) Diet
  Arms: Low-Fat/Low-Sugar (LF/LS) Diet

SUMMARY:
In this randomized, single-blinded basic research study, healthy normal-weight human participants are exposed to a high-fat/high-sugar (HF/HS) snack or a low-fat/low-sugar (LF/LS) snack twice a day for eight weeks in addition to their regular diet. All participants are tested at baseline, after 4 weeks and after 8 weeks of dietary intervention.

At all time points the investigators acquire the following parameters:

* Body weight and composition,
* Blood parameters to control for metabolic changes,
* Visual analog scales (hunger, satiety, tiredness, etc.),
* Fat and sugar concentration preference,
* Functional Magnetic Resonance Imaging (fMRI) during a learning and a gustatory perception task.

The investigators hypothesize that the habitual consumption of a small HF/HS snack will reduce the preference for low-fat concentrations and will have an impact on brain response to the anticipation and consumption of palatable food. Moreover, the investigators hypothesize, that HF/HS diet will have an impact neuronal encoding of learning independent of food cues. The investigators expect these alterations independent of body weight gain suggesting a direct effect of HF/HS diet on neuronal circuits.

DETAILED DESCRIPTION:
In this randomized, single-blinded basic research study, healthy normal-weight human participants are exposed to a high-fat/high-sugar (HF/HS) snack or a low-fat/low-sugar (LF/LS) snack twice a day for eight weeks in addition to their regular diet. The investigators test the effect of this dietary intervention on body weight, metabolic parameters such as insulin sensitivity, blood cholesterol and triglycerides, the preference of fat and sugar taste, the brain response to milkshake anticipation and consumption, and as the neuronal coding of prediction error learning. Here, all participants are tested at baseline, after 4 weeks and after 8 weeks of dietary intervention using behavioral tasks, fMRI and blood sampling. The investigators hypothesize that the habitual consumption of a small HF/HS snack will reduce the preference for low-fat concentrations and impact brain response to the anticipation and consumption of palatable food. Moreover, the investigators hypothesize, that HF/HS diet will have an impact neuronal encoding of learning independent of food cues. The investigators expect these alterations independent of body weight gain suggesting a direct effect of HF/HS diet on neuronal circuits.

ELIGIBILITY:
Inclusion Criteria:

* right handed
* non-smoker (for the last 1 year not smoked more than 2 cigarettes per month)
* Body Mass Index between 20-27 kg/m2 (healthy weight)

Exclusion Criteria:

1. serious or unstable medical illness (e.g., cancer);
2. past or current history of alcoholism or consistent drug use;
3. current and history of major psychiatric illness as defined by the DSM-IV (Diagnostic and Statistical Manual) criteria including eating disorders,
4. medications that affect alertness (e.g., barbiturates, benzodiazepines, chloral hydrate, haloperidol, lithium, carbamazepine, phenytoin, etc.) and any psychoactive drugs or anti-obesity agents;
5. history of major head trauma with loss of consciousness;
6. ongoing pregnancy;
7. known taste or smell dysfunction;
8. a diagnosis of diabetes;
9. any known food allergy, certain food sensitivities (lactose);
10. pregnant or nursing women,
11. history of metalworking, injury with shrapnel or metal slivers, and major surgery;
12. history of pacemaker or neurostimulator implantation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

PRIMARY OUTCOMES:
Change in fat taste preference after 8-weeks dietary intervention | Preference (wanting and liking) for different fat and sugar concentrations was assessed at baseline and after the 8-weeks intervention.
  In the fat and sugar concentration preference task, the preference and perception are evaluated using a series of puddings with varying fat content (0%, 3.1%, 6.9%, and 15.6 %), and sugar concentration using apple juice with varying sucrose content (0 M, 0.1 M, 0.56 M, and 1 M). Each pudding and juice concentration is tested 12 times and the average is calculated. "Wanting" and "Liking" are assessed for all concentrations and the change between baseline and the post-intervention is assessed in both HF/HS and LF/LS groups.
Change brain response to milkshake anticipation and milkshake consumption after 8-weeks dietary intervention | BOLD (blood oxygen level-dependent) response to milkshake anticipation and consumption was assessed at baseline and after the 8-weeks intervention.
  To test the effect of the dietary intervention on brain responses to milkshake anticipation (milkshake predicting cue) and consumption (milkshake delivery), the investigators performed a gustatory perception task. The BOLD response while milkshake cue presentation and milkshake delivery was compared between baseline and postintervention and compared between groups.
Change in neuronal encoding of prediction error processing after 8-weeks dietary intervention. | BOLD response related to choice prediction error was assessed at baseline and after 8 weeks of intervention. (http://www.vislab.ucl.ac.uk/Cogent/index.html).For further analysis, the investigators calculated the average rating across the total 12.
  A short version of the sensory learning task as described in detail by Iglesias et al. (2019) was performed to assess associative learning independent of food rewards, while undergoing fMRI. Within this model, the investigators computed the (signed) adaptive precision error relating to the precision-weighted choice prediction error about visual outcome, that is, the product of choice prediction error (a) and the adaptive learning rate (b). The investigators tested the BOLD response related to choice prediction error and compared it between baseline and post-intervention and between the HF/HS and LF/LS group.

CONTACTS AND LOCATIONS:
Overall Officials: Jens C Bruening, MD, Study Director — Max Planck Institute for Metabolism Research; Dana M Small, PhD, Principal Investigator — Yale University; Marc Tittgemeyer, PhD, Principal Investigator — Max Planck Institute for Metabolism Research